CLINICAL TRIAL: NCT03964077
Title: Turkish Version of the Neurogenic Bladder Symptom Score Questionnaire: a Cross-cultural Adaptation, Reliability and Validity Study
Status: Completed | Type: Observational
Sponsor: Gaziosmanpasa Research and Education Hospital (Other Government)
Responsible Party: Principal Investigator, Mehmet Akif GÜLER, Principal Investigator, Gaziosmanpasa Research and Education Hospital
Other Study IDs: GaziosmanpasaTREH6
Record Dates: First submitted 2019-05-22; First posted 2019-05-28 (Actual); Last update posted 2020-01-28 (Actual); Status verified 2020-01

CONDITIONS: Spinal Cord Injuries
Keywords: Neurogenic Bladder; Quality of life; Spinal Cord Injury
MeSH Terms: conditions — Spinal Cord Injuries; Urinary Bladder, Neurogenic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Neurogenic Bladder Symptom Score Questionnaire — Neurogenic Bladder Symptom Score Questionnaire is a self-reported 24 item questionnaire.

SUMMARY:
Turkish version of the Neurogenic Bladder Symptom Score questionnaire: a cross-cultural adaptation, reliability and validity study

DETAILED DESCRIPTION:
Turkish version of the Neurogenic Bladder Symptom Score questionnaire: a cross-cultural adaptation, reliability and validity study in spinal cord patients.

ELIGIBILITY:
Inclusion Criteria:

* Spinal cord injury patients
* aged > 18 years old

Exclusion Criteria:

* spinal shock patients
* urinary tract operation in the last month
* Quality of life changes in the last month
* urinary tract infections in the last month
* bladder management changes or drug changes in the last month

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 70 spinal cord injury patients
Sampling Method: Probability Sample
Enrollment: 102 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2020-01-27 (Actual); Study Completion 2020-01-27 (Actual)

PRIMARY OUTCOMES:
Life quality: Short-form 36 | 4 months
  The quality of life of the patients will be determined using Short-form 36. The self-reported questionnaire includes 8 domains (using algorithms) (0-100 points). Higher scores show poorer quality of life.
Neurogenic Bladder Symptom Score Questionnaire | 4 months
  Neurogenic Bladder Symptom Score Questionnaire is a 24 item self-reported questionnaire(0-74 points). The questionnaire includes 4 subgroups; incontinence (0-29 points), storage&voiding (0-22 points) and consequences (0-23 points). Higher the score, the greater the severity of the symptoms.
The King's Health Questionnaire | 4 months
  The King's Health Questionnaire (KHQ) is one of the most widely used for assessing QOL in patients with urinary inkontinence.The KHQ consists of two parts and 32 items [7]. The first part (21 items) contains two single-item questions that address General Health Perception and Incontinence Impact and the following seven multi-item domains: Role, Physical, and Social Limitations, Limitations in Personal Relationship, Emotional Problems, Sleep and Energy Disturbances associated with UI, and Severity Measures for UI. The second part has an 11-item Symptom Severity Scale (SSS) that assesses the presence and severity of urinary symptoms. While the entire SSS is scored from 0 (best) to 30 (worst), the minimum possible score is 0 (best health) and the maximum possible score is 100 (worst health) for all other KHQ domains.

CONTACTS AND LOCATIONS:
Locations (1):
- Mehmet Akif Guler, Istanbul, İ̇stanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Guler MA, Dogan D, Yilmaz Yalcinkaya E. Validity and reliability of the Turkish version of the neurogenic bladder symptom score. Disabil Rehabil. 2022 Jun;44(12):2889-2895. doi: 10.1080/09638288.2020.1846216. Epub 2020 Nov 24. PMID 33232613